CLINICAL TRIAL: NCT02209714
Title: A Single Increasing Dose Safety, Tolerability and Pharmacodynamics (Citric Acid Challenge) Study After Oral Administration of BIIF 1149 BS (Single Doses as Tablets: 40, 65, 100 mg) in Healthy Male Volunteers (Randomised, Double-blind Within Each Dose Group, Placebo-controlled, Parallel Groups)
Brief Title: Safety, Tolerability and Pharmacodynamics After Oral Administration of BIIF 1149 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1157.4
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BIIF 1149 BS (Experimental)
  Interventions: Drug: BIIF 1149 BS
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIF 1149 BS
  Arms: BIIF 1149 BS
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to obtain information about the safety and tolerability of BIIF 1149 BS45 (single dose: 40, 65, 100 mg), to determine the pharmacologically active dose (range) by performing a citric acid challenge test and to obtain preliminary pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, based on a complete medical examination
* Age range from 21 to 50 years
* +/- 20 % of their normal weight (Broca-Index)
* Written informed consent

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with known history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections (especially respiratory infections, cough)
* Volunteers with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Volunteers who have taken a drug with a long half-life (≥ 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Volunteers who received any other drugs which might influence the results of the study during the week prior to the start of the study
* Volunteers who have participated in another study with an investigational drug within the last 2 months preceding this study
* Volunteers who smoke more than 10 cigarettes (or equivalent) per day
* Volunteers who are not able to refrain from smoking on study days
* Volunteers who drink more than 40 g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who are participated in excessive physical activities (e.g. competitive sports) during the last week before the study
* Volunteers who have donated blood (≥ 100 ml) within the last four weeks

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1999-11; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant changes in vital functions (blood pressure, pulse rate) | up to 8 days after last drug administration
Number of patients with clinically relevant changes in electrocardiogram (ECG) | up to 8 days after last drug administration
Number of patients with clinically relevant changes in laboratory parameters | up to 8 days after last drug administration
Number of patients with adverse events | up to 8 days after last drug administration

SECONDARY OUTCOMES:
Maximum drug plasma concentration (Cmax) | up to 360 hours after drug administration
Time to reach maximum drug concentration (tmax) | up to 360 hours after drug administration
Total area under the plasma drug concentration-time curve (AUC) for several time points | up to 360 hours after drug administration
Terminal half-life (t1/2) | up to 360 hours after drug administration
Mean residence time (MRT) | up to 360 hours after drug administration
Total clearance after oral administration (CLtot/f) | up to 360 hours after drug administration
Amount of drug excreted in urine (Ae) | up to 360 hours after drug administration
Measurement of pharmacodynamic activity | Screening, at least 15 days after first administration
  Citric acid challenge
Volume of Distribution during terminal phase after oral administration (Vz/F) | up to 360 hours after drug administration
Renal clearance in the time interval form 0 to x h (Clren0-xh) | up to 360 hours after drug administration